CLINICAL TRIAL: NCT00559975
Title: A Phase 1, Randomized, Controlled, Observer-Blinded, Dose Escalation Study of the Safety, Tolerability and Immunogenicity of a Single Dose of Adjuvanted Influenza Vaccine Combined With CpG7909 in Healthy Adults
Brief Title: Safety, Tolerability, Immunogenicity And CPG Dosage Finding Study of Novartis CpG Adjuvanted Flu Vaccine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis (Industry)
Collaborators: Novartis Vaccines (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: V95P1
Record Dates: First submitted 2007-11-16; First posted 2007-11-19 (Estimated); Last update posted 2009-11-05 (Estimated); Status verified 2009-11

CONDITIONS: Influenza Infection
Keywords: Adjuvanted Influenza Vaccine
MeSH Terms: interventions — ProMune

STUDY DESIGN:
Who Masked: Participant

ARMS (5):
- 1 (Active Comparator)
  Interventions: Biological: Subunit influenza vaccine
- 2 (Active Comparator)
  Interventions: Biological: Adjuvanted influenza vaccine
- 3 (Experimental)
  Interventions: Biological: Adjuvanted influenza vaccine combined with CpG7909
- 4 (Experimental)
  Interventions: Biological: Adjuvanted influenza vaccine combine with CpG7909
- 5 (Experimental)
  Interventions: Biological: Adjuvanted influenza vaccine combine with CpG7909

INTERVENTIONS:
Biological: Subunit influenza vaccine — 0.5 mL single dose vaccine
  Arms: 1
Biological: Adjuvanted influenza vaccine — 0.5 mL single dose vaccine
  Arms: 2
Biological: Adjuvanted influenza vaccine combined with CpG7909 — 0.5 ml influenza vaccine combined with 10 mcg of CpG7909
  Arms: 3
Biological: Adjuvanted influenza vaccine combine with CpG7909 — 0.5 mL single dose vaccine combined with 30 mcg of CpG7909
  Arms: 4
Biological: Adjuvanted influenza vaccine combine with CpG7909 — 0.5 mL single dose vaccine combined with 100 mcg of CpG7909
  Arms: 5

SUMMARY:
To evaluate the safety and tolerability of the an adjuvanted influenza vaccine combined with CpG7909 at three different doses of CpG 7909 as a single intramuscular (IM) administration in healthy adults. Safety will be assessed by observation of symptoms, physical examination findings and laboratory safety testing.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects aged 18 to ≤40 years

Exclusion Criteria:

* Any serious disease, hypersensitivity to egg or vaccine components, neurological symptoms or positive antibody test against dsDNA, RF, ANA or thyroid.
* Abnormal TSH from blood samples collected during the screening visit;

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2007-10; Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Measures of humoral immunogenicity for each antigen | 22 days

SECONDARY OUTCOMES:
Measures of vaccine-induced B and T cell immune responses | 72 hours
Measure of alterated biomarkers and measure of safety | 72 hours

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Vaccines, Study Chair — Novartis Vaccines
Locations (1):
- Institute for Pharmacokinetic and Analytical Studies, Ligornetto, Switzerland